CLINICAL TRIAL: NCT05195554
Title: Effectiveness of a Psycho-educational Intervention for People With Suicidal Conduct in the Prison Environment. N'VIU Project: a Randomized Control Trial
Brief Title: A Psycho-educational Intervention for People With Suicidal in Prisons
Acronym: N'VIU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Consorci Hospitalari de Vic (Other)
Collaborators: Government of Catalonia (Unknown)
Responsible Party: Principal Investigator, Dr. Pere Roura-Poch, Head of epidemiology, Consorci Hospitalari de Vic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021059
Record Dates: First submitted 2021-12-30; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Suicide
Keywords: suicide; suicide behaviour; suicide prevention; prison environment; psychoeducational intervention; randomized controlled trial
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: The study design is a multicentric, randomized, controlled trial with two parallel groups, with blind assessment of the response variables, with a 12-months of follow-up.
Who Masked: Outcomes Assessor
Masking Description: Blind assessment of the response variables.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention groups will involve a psycho-educational intervention and will consist of between 10 and 12 people led by two professionals, one of whom must be a psychologist, while the other may be any professional in the center (usually social workers).
  Interventions: Other: Psycho-educational intervention
- Control group (No Intervention): Participants in the control group will receive information on suicide and advice if the suicidal ideation increases.

INTERVENTIONS:
Other: Psycho-educational intervention — Psycho-educational intervention will consist of between 10 and 12 people led by two professionals.
  Arms: Intervention group

SUMMARY:
This study has been designed as a multicentric, randomized, two parallel-group, controlled trial. The study population will be male and female inmates of nine prisons of Catalonia (Spain). The primary outcome will be the total number of suicidal behaviours for 12 months of follow-up. This project aims to assess the effectiveness of a psycho-educational intervention on reducing the number of suicidal behaviours in the prison environment. If positive, the prison community will have a new tool to curb suicide in prisons.

DETAILED DESCRIPTION:
Background: Suicide rates are higher in the prison environment than in the general population. Prevention involves strategies to promote mental health, early diagnosis, treatment and identification of precipitating factors. The aim of this study is to evaluate the effectiveness of a psychoeducational group intervention performed by rehabilitation professionals to decrease the number of suicidal behaviors in the penitentiary environment.

Methods: This study has been designed as a multicentric, randomized, two parallel-group, controlled trial. The study population will be male and female inmates of nine prisons of Catalonia (Spain). The primary outcome will be the total number of suicidal behaviours for 12 months of follow-up. Secondary outcomes will be suicide risk evaluated with the International Neuropsychiatric Interview (MINI); the severity of suicidal ideations assessed with the Columbia-Suicide Severity Rating Scale (C-SSRS), the presence of depressive and anxiety symptoms [Hamilton Depression Rating Scale (HDRS) and Hamilton Anxiety Rating Scale (HARS)] and health-related quality of life (EQ-5D). Other variables will be clinical and socio-demographic. Intervention will consist of 17 psychoeducation sessions for the intervention group and information on suicide for the control group.

Conclusions: This project aims to assess the effectiveness of a psycho-educational intervention on reducing the number of suicidal behaviours in the prison environment. If positive, the prison community will have a new tool to curb suicide in prisons.

ELIGIBILITY:
Inclusion Criteria:

- Participants who have presented some kind of suicidal or high-risk behavior in the criterion of self-directed violence according to the RisCanvi*.

Exclusion Criteria:

* Decompensation of severe mental disorder
* Intellectual disability
* Cognitive impairment.
* Isolation

  * RisCanvi is an instrument used by penitentiary professionals, based on the individualized and structured assessment of a set of pre-established variables, in order to manage the probabilities of increased and decreased risk of prison inmates for further episodes of violent behavior. The full RisCanvi scale consists of 43 risk factors grouped in the following areas: criminological, personal and biographical, social, family, clinical, and personality. These 43 factors are added to the assessment of the future risk of the emergence of four behaviors: self-directed violence, intra-institutional violence, repeat violence, and prison-breaking).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Total number of suicidal behaviours | 12 months
  The primary outcome will be the total number of suicidal behaviours -which includes both suicide attempts and suicides- registered during the first year after being included in the study.

SECONDARY OUTCOMES:
Suicide risk | 12 months
  This risk will be evaluated with the International Neuropsychiatric Interview (MINI). The MINI is a structured diagnostic interview, of short duration, with six yes or no questions. It allows for a score between 0 and 35, with 1-5 corresponding to a slight suicide risk, 6-9 moderate and 10 high.
Severity of suicidal ideation | 12 months
  The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess the seriousness of the suicidal ideation. C-SSRS will be used to assess the seriousness of the suicidal ideation, included four constructs: 1) the severity of ideation, with a subscale that evaluates 5 types of increasing gravity (from 1: wish to be dead; to 5: active suicidal ideation with specific plan and intent); 2) intensity of ideation, consisting of 5 elements -frequency, duration, controllability, deterrents, reasons for ideation- each with a subscale from either 0 to 5 or 1 to 5. 3) suicidal behavior, with a subscale that evaluates with a nominal scale actual, interrupted and aborted attempts, preparatory acts and non-suicidal self-destructive conduct; and 4) lethality of the suicide attempt, which evaluates with an ordinal scale of 6 points (from 0: there is no physical damage to 5: death.
Depression | 12 months
  We will evaluate the presence of depressive symptoms with the Hamilton Depression Rating Scale (HDRS). The scale provides a global score of severity of the depression between 0 and 52. The cutting points recommended by the National Institute for Health and Care Excellence (NICE) guide are: 0-7: non-depression; 8-13: light depression; 14-18: moderate depression; 19-22: severe depression, and ≥23: very severe depression.
Anxiety | 12 months
  To evaluate the presence of anxiety symptoms, we will use the Hamilton Anxiety Rating Scale (HARS), a hetero-administered scale that aims to assess the intensity of anxiety. It consists of 14 items that evaluate the mental, physical and behavioral aspects of anxiety. The time frame is the previous 3 days on all items except the last. It provides a global measure of anxiety obtained by adding the score obtained in each item, with 0-5 indicating non-anxiety; 6-14 mild anxiety; and ≥15 moderate/severe anxiety. There is a validated Spanish version.
Quality of life (QOL) | 12 months
  This will be measured through the EuroQoL-5D Health Questionary (EQ-5D), a self-applied questionnaire consisting of two parts: the first assesses 5 dimensions: mobility, personal care, everyday activities, pain/disease and anxiety/depression. For each dimension, three states are described: absence of problems (1 point), moderate problems (2 points) or severe problems (3 points). The second part is visual analogue scale represented by a graduated vertical line from 0 (worst imaginary state of health) to 100 (best imagined state of health). It is validated in Catalan.

CONTACTS AND LOCATIONS:
Overall Officials: Quintí Foguet-Boreu, MD,PhD, Principal Investigator — Consorci Hospitalari de Vic
Locations (1):
- Vic University Hospital, Vic, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suicide worldwide in 2019: global health estimates. Geneva: World Health Organization; 2021. Available at: https://www.who.int/teams/mental-health-and-substance-use/data-research/suicide-data. Accessed 10 December 2021.
- [Background] Ministerio del Interior. Mortalidad en Instituciones Penitenciària s (II.PP.) Año 2017. Boletín epidemiológico de Instituciones Penitenciària. 2019; 24 (2).
- [Background] Department of Justice. Penitentiary services. Statistics data 2018. Available at: http://justicia.gencat.cat/ca/departament/Estadistiques/serveis_penitenciaris. Accessed 10 December 2021.
- [Background] World Health Organization. Preventing suicide in jails and prisons. Geneve: WHO; 2007.
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Ferrando L, Bobes J, Gibert M, Soto M, Soto O. M.I.N.I. Mini International Neuropsychiatric Interview. Versión en español 5.0.0.DSM-IV. Instituto IAP, Madrid, 1998
- [Result] Zhong S, Senior M, Yu R, Perry A, Hawton K, Shaw J, Fazel S. Risk factors for suicide in prisons: a systematic review and meta-analysis. Lancet Public Health. 2021 Mar;6(3):e164-e174. doi: 10.1016/S2468-2667(20)30233-4. Epub 2021 Feb 10. PMID 33577780
- [Result] Cramer RJ, Wechsler HJ, Miller SL, Yenne E. Suicide Prevention in Correctional Settings: Current Standards and Recommendations for Research, Prevention, and Training. J Correct Health Care. 2017 Jul;23(3):313-328. doi: 10.1177/1078345817716162. Epub 2017 Jun 28. PMID 28656789
- [Result] Pratt D, Tarrier N, Dunn G, Awenat Y, Shaw J, Ulph F, Gooding P. Cognitive-behavioural suicide prevention for male prisoners: a pilot randomized controlled trial. Psychol Med. 2015 Dec;45(16):3441-51. doi: 10.1017/S0033291715001348. Epub 2015 Jul 13. PMID 26165919
- [Result] Kazis LE, Anderson JJ, Meenan RF. Effect sizes for interpreting changes in health status. Med Care. 1989 Mar;27(3 Suppl):S178-89. doi: 10.1097/00005650-198903001-00015. PMID 2646488
- [Result] Leidenfrost CM, Schoelerman RM, Maher M, Antonius D. The development and efficacy of a group intervention program for individuals with serious mental illness in jail. Int J Law Psychiatry. 2017 Sep-Oct;54:98-106. doi: 10.1016/j.ijlp.2017.06.004. Epub 2017 Jun 24. PMID 28655427
- [Result] Winicov N. A systematic review of behavioral health interventions for suicidal and self-harming individuals in prisons and jails. Heliyon. 2019 Sep 6;5(9):e02379. doi: 10.1016/j.heliyon.2019.e02379. eCollection 2019 Sep. PMID 31517115
- [Result] Johnson JE, Stout RL, Miller TR, Zlotnick C, Cerbo LA, Andrade JT, Nargiso J, Bonner J, Wiltsey-Stirman S. Randomized cost-effectiveness trial of group interpersonal psychotherapy (IPT) for prisoners with major depression. J Consult Clin Psychol. 2019 Apr;87(4):392-406. doi: 10.1037/ccp0000379. Epub 2019 Feb 4. PMID 30714749
- [Result] Eck M, Scouflaire T, Debien C, Amad A, Sannier O, Chan Chee C, Thomas P, Vaiva G, Fovet T. [Suicide in prison: Epidemiology and prevention]. Presse Med. 2019 Jan;48(1 Pt 1):46-54. doi: 10.1016/j.lpm.2018.11.009. Epub 2019 Jan 23. French. PMID 30685227